CLINICAL TRIAL: NCT05113004
Title: NEw Clinical Endpoints in Patients With Primary Sjögren's Syndrome (pSS): an Interventional Trial Based on stratifYing Patients
Brief Title: New Clinical End-points in Patients With Primary Sjögren's Syndrome
Acronym: NECESSITY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP190131
Record Dates: First submitted 2021-11-02; First posted 2021-11-09 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Primary Sjögren's Syndrome (pSS)
Keywords: dry eye; Oral Dryness and Saliva Altered; Eular Sjögren Syndrome Disease Activity index; Primary Sjögrens's syndrome
MeSH Terms: conditions — Dry Eye Syndromes; Xerostomia | interventions — Hydroxychloroquine; Leflunomide; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, randomized, double blinded
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm 1 (Placebo Comparator): Cohort 1 : Patients with High levels of symptoms and low disease activity receive :
  Placebo of Leflunomide 20mg/d Placebo of Mycophenolate mofetil 2000mg/d Placebo of hydroxychloroquine 400mg/d
  Interventions: Drug: Placebo of Hydroxychloroquine 400mg/d; Drug: Placebo of Leflunomide 20mg/d; Drug: Placebo of Mycophenolate mofetil 2000mg/d
- Arm 2 (Other): Cohort 1 : Patients with High levels of symptoms and low disease activity receive :
  Leflunomide 20mg/d hydroxychloroquine 400mg/d Placebo of Mycophenolate mofetil 2000 mg/d
  Interventions: Drug: Hydroxychloroquine 400mg/d; Drug: Leflunomide 20mg/d; Drug: Placebo of Mycophenolate mofetil 2000mg/d
- Arm 3 (Other): Cohort 1 : Patients with High levels of symptoms and low disease activity receive :
  Placebo of Leflunomide 20mg/d Mycophenolate mofetil 2000mg/d hydroxychloroquine 400mg/d
  Interventions: Drug: Hydroxychloroquine 400mg/d; Drug: Mycophenolate mofetil 2000mg/d; Drug: Placebo of Leflunomide 20mg/d
- Arm 4 (Placebo Comparator): Cohorte 2 :Patients with moderate or hight activity, regardless of level of symptoms, they receive :
  Placebo of Leflunomide 20mg/d Placebo of Mycophenolate mofetil 2000mg/d Placebo of hydroxychloroquine 400mg/d
  Interventions: Drug: Placebo of Hydroxychloroquine 400mg/d; Drug: Placebo of Leflunomide 20mg/d; Drug: Placebo of Mycophenolate mofetil 2000mg/d
- Arm 5 (Other): Cohorte 2 :Patients with moderate or hight activity, regardless of level of symptoms, they receive :
  Leflunomide 20mg/d hydroxychloroquine 400mg/d Placebo of Mycophenolate mofetil 2000 mg/d
  Interventions: Drug: Hydroxychloroquine 400mg/d; Drug: Leflunomide 20mg/d; Drug: Placebo of Mycophenolate mofetil 2000mg/d
- Arm 6 (Other): Cohorte 2 :Patients with moderate or hight activity, regardless of level of symptoms, they receive :
  Placebo of Leflunomide 20mg/d Mycophenolate mofetil 2000mg/d hydroxychloroquine 400mg/d
  Interventions: Drug: Hydroxychloroquine 400mg/d; Drug: Leflunomide 20mg/d; Drug: Placebo of Leflunomide 20mg/d

INTERVENTIONS:
Drug: Hydroxychloroquine 400mg/d — Hydroxychloroquine (HCQ) is a 4-aminoquinoline belonging to the group of antimalarial agents. Its immunomodulatory activity on B-cells has mainly been attributed to its inhibition of antigen presentation, cytokine production, and recently on Toll-like receptor signaling and IFN secretion that drives B cell activation.
  Arms: Arm 2; Arm 3; Arm 5; Arm 6
Drug: Leflunomide 20mg/d — Leflunomide (LEF) is a derivative of isoxazole and is converted into an active metabolite which blocks de novo synthesis of pyrimidines in activated T lymphocytes, thereby inhibiting T cell proliferation and consequently T cell-dependent B cell formation of autoantibodies.
  Arms: Arm 2; Arm 5; Arm 6
Drug: Mycophenolate mofetil 2000mg/d — Mycophenolate mofetil (MMF) is a morpholinoethyl ester of mycophenolic acid which blocks proliferation of lymphocytes by inhibiting the de novo pathway of purine biosynthesis (Allison, 2000).
  Arms: Arm 3
Drug: Placebo of Hydroxychloroquine 400mg/d — Placebo of Hydroxychloroquine (HCQ) is a 4-aminoquinoline belonging to the group of antimalarial agents. Its immunomodulatory activity on B-cells has mainly been attributed to its inhibition of antigen presentation, cytokine production, and recently on Toll-like receptor signaling and IFN secretion that drives B cell activation.
  Arms: Arm 1; Arm 4
Drug: Placebo of Leflunomide 20mg/d — Placebo of Leflunomide (LEF) is a derivative of isoxazole and is converted into an active metabolite which blocks de novo synthesis of pyrimidines in activated T lymphocytes, thereby inhibiting T cell proliferation
  Arms: Arm 1; Arm 3; Arm 4; Arm 6
Drug: Placebo of Mycophenolate mofetil 2000mg/d — Placebo of Mycophenolate mofetil (MMF) is a morpholinoethyl ester of mycophenolic acid which blocks proliferation of lymphocytes by inhibiting the de novo pathway of purine biosynthesis (Allison, 2000).
  Arms: Arm 1; Arm 2; Arm 4; Arm 5

SUMMARY:
There are no approved treatments for pSS and the clinical endpoints currently used in clinical trials are inadequate to capture all aspects of the disease that should be evaluated in clinical trials. The newly developed composite endpoint: Sjögren's Tool for Assessing Response to treatment (STAR) will allow a more specific and meaningful assessment of treatment efficacy in pSS.

Because of the heterogeneity of the disease and of the central role of the interplay between B- and T-cells in the pathogenesis, it is worth to evaluate combination of conventional synthetic immunomodulatory drugs targeting both B- and T-cells.

DETAILED DESCRIPTION:
Primary Sjögren's syndrome (pSS) is a systemic autoimmune disease with a female-to-male predominance of 9:1 and a peak incidence at 50 years of age. It is characterized by chronic inflammation and subsequent destruction of exocrine glands, mainly lacrimal and salivary glands, with ocular and oral dryness. Patients also experience joint pain and extreme fatigue. In 20-40% of patients, the inflammatory process extends beyond the exocrine glands and patients experience systemic extra glandular manifestations, with 5-10% developing B-cell lymphoma.

Two populations of pSS patients can be defined. Patients with dryness, fatigue, pain and low systemic activity present no or limited long-term extraglandular damage but they have a profoundly reduced quality of life with marked anxiety, depression, and social isolation (Rischmueller 2016)(Meijer, 2009). Patients with high systemic activity have important long-term damage and bad prognosis. To date, there are no approved disease-modifying treatments.

Current clinical outcome assessment (COA) tools in pSS have shown important weaknesses (e.g. high placebo response rate) which may hamper demonstration of therapeutic benefit. A novel COA called STAR has recently been developed by the NECESSITY consortium (funded by the Innovative Medicines Initiative) and should allow the identification of new therapeutic options for both patient populations.

the investigator aim to demonstrate, thanks to the new STAR outcome measure, efficacy of a combination therapy targeting both B- and T-cells in pSS patients.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1
* Having given written informed consent prior to undertaking any study-related procedures.
* Patients with pSS according to ACR/EULAR 2016 criteria or AECG 2002 criteria
* With a high level of symptoms (ESSPRI ≥ 5) and low systemic disease activity (ESSDAI < 5).
* Negative pregnancy test (serum at screening)
* Use highly reliable contraception during research treatment from the screening and for two years after stopping treatment.
* Cohort 2
* Having given written informed consent prior to undertaking any study-related procedures.
* Patients with pSS according to ACR/EULAR 2016 criteria or AECG 2002 criteria
* With moderate/high systemic disease activity, as defined by ESSDAI ≥ 5.
* Negative pregnancy test (serum at screening)
* Use highly reliable contraception during research treatment from the screening and for two years after stopping treatment

Exclusion Criteria:

* For both cohorts:
* Age < 18 years
* Pregnant or breastfeeding women or women wanted to conceive either during or within two years after the end of the treatment period
* Women of childbearing potential not using highly effective methods of contraception (as defined in section 6.3)
* Participation in another interventional trial
* Contra-indication to HCQ: pre-existing retinopathy, hypersensitivity to HCQ or to any of the excipients of the specialty used
* Contra-indication to MMF: hypersensitivity to mycophenolate mofetil, acid mycophenolic, mycophenolate sodium or to any of the excipients of the specialty used
* Contra-indication tor LEF: hypersensitivity to the active substance, the main active metabolite teriflunomide or to any excipients of the specialty used.
* Concomitant treatment with corticosteroids more than 10 mg/day of prednisone equivalent at screening or inclusion (randomisation)
* Concomitant treatment with other immunomodulators including methotrexate, azathioprine, cyclophosphamide, cyclosporine and tacrolimus
* Previous treatment with HCQ, LEF, MMF in the last 3 months
* Previous treatment with rituximab, other B-cell targeted biologic therapy or cyclophosphamide in the last 6 months
* Previous treatment with anti-TNF, abatacept, tocilizumab or belimumab or any other biologic in the setting of a past clinical trial in the last 3 months
* Severe life-threatening systemic involvement requiring cyclophosphamide or high dose corticosteroids, or any drug considered as an exclusion criteria
* Impairment of other severe immunodeficiency states
* Patients with active malignancy or history of malignancy within the last 5 years except non-melanoma skin cancer
* Patients with history of gastrointestinal tract ulceration, hemorrhage and perforation
* Patients with history of cardiomyopathy
* Patients with known hereditary deficiency of hypoxanthine-guanine phosphoribosyl-transferase (HGPRT) such as Lesch-Nyhan and Kelley-Seegmiller syndrome
* Serious infection in the past month
* Evidence of active tuberculosis infection
* Active HCV (positive PCR)
* Active HBV infection (positivity for HBS antigen, or positivity for anti-HBC antibody without any HBS antigen)
* HIV infection (positive serology)
* Positive SARS-Cov2 PCR (if vaccinated for COVID-19, no PCR is required; if history of COVID-19 infection, positive serology is sufficient)
* Cytopenia defined as neutrophils < 1.0 G/L, lymphocytes < 0.5 G/L, Hb < 10 g/dl or platelets < 100 G/L
* Moderate to severe renal insufficiency (GFR < 30 ml/min)
* Severe hypogammaglobulinemia defined as gamma globulins or IgG < 5 g/l Reduced hepatic function: AST or ALT > 2x ULN (re-testing is allowed, see section 5.10)
* Prolonged ECG's corrected QT interval (>500 ms)
* Known history of maculopathy
* Patients will be informed of the risk of alcohol consumption and will be recommended to avoid alcohol during the entire study
* Not affiliated to a social security regime (specific for France)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Cohort 1. Proportion of patients achieving a response according to preliminary STAR at week 24 between each active treatment arm and placebo arm. | During the 24 weeks of the trials
Cohort 2. Proportion of patients achieving a response according to preliminary STAR at week 24 between each active treatment arm and placebo arm. | During the 24 weeks of the trials

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Valérie Devauchelle, Brest
  - Eric Hachulla, Lille
  - Jacques Morel, Montpellier
  - Véronique Le Guern, Paris
  - Jacques-Eric Gottenberg, Strasbourg
  - Christophe Richez, Talence
  - Raphaele Seror, Le Kremlin-Bicêtre, Île-de-France Region